CLINICAL TRIAL: NCT01567215
Title: Treatment of Granuloma Umbilical in Newborn Babies - Comparison of Treatment With Silver Nitrate Versus Alcohol Swaps Versus Steroid Creme Group IV
Brief Title: Treatment of Granuloma Umbilical in Newborn Babies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pernille Pedersen (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor-Investigator, Pernille Pedersen, Doctor Pernille Pedersen, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201201; 2011-005300-15 (EudraCT Number)
Record Dates: First submitted 2012-03-22; First posted 2012-03-30 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Fetus or Newborn Affected by Condition of Umbilical Cord
Keywords: granuloma umbilical
MeSH Terms: interventions — Silver Nitrate; Steroids; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Granuloma (Experimental)
  Interventions: Procedure: silver nitrate; Drug: Steroids; Procedure: alcohol

INTERVENTIONS:
Procedure: silver nitrate — Application 1 - 2 times a week for 3 - 4 weeks
  Other Names: Product ATC code D08AL01
Drug: Steroids — Dermovate creme group IV steroid. Application 2 times a day for 3 weeks or less if the granuloma disappears.
  Other Names: Clobetasolpropionat 0,5 mg/g; ATC kode D07AD01
Procedure: alcohol — Alcohol swabs 82% ethanol. Application 6 - 8 times a day, each time the parents change the diaper. Treatment for 3 weeks or less if the granuloma disappears.
  Other Names: 82% ethanol

SUMMARY:
The investigators want to show that steroid creme and even better alcohol swaps are just as effective or equal to the current treatment with silver nitrate of granuloma umbilical in newborns.

DETAILED DESCRIPTION:
The change of treatment will make it possible for parents to treat the children themselves at home, whereas treatment with silver nitrate only is an in hospital regimen.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age more than 37 weeks
* More than 3 weeks old baby
* Granuloma umbilical diagnosed by a pediatrician
* No infections due to the umbilicus
* Parents do understand and speak danish

Exclusion Criteria:

* Gestational age less than 37 weeks
* Less than 3 weeks old baby
* Granuloma umbilical not diagnosed by a pediatrician
* Infections due to the umbilicus
* Parents do not understand or speak Danish

Ages: 3 Weeks to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Is alcohol swabs and steroid creme as effective as lapis in treatment of granuloma umbilica? | 2 years
  Change current treatment of Grauloma Umbilical. Show that alcohol swaps or steroid creme group IV are just as effective as current treatment of granuloma umbilica with silver nitrate.

SECONDARY OUTCOMES:
Change of treatment of granuloma umbilical in hospitals by professionals to treatment at home by parents | 2 years
  Change current treatment of granuloma umbilica with silver nitrate at hospitals to treatment at home by parents.

OTHER OUTCOMES:
Avoid side effects by changing treatment of granuloma umbilical | 2 years
  Severe side effect as skinburns is seen by using silver nitrate treating granuloma umbilica, using alcohol swabs or steroid creme less side effects are seen?

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Pedersen, Doctor, Principal Investigator — Hvidovre University Hospital, Childrens apartement
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Kettegård Alle 31, Hvidovre
  - Hvidovre University Hospital, Hvidovre, Kettegård Alle 30

REFERENCES:
- [Background] Nagar H. Umbilical granuloma: a new approach to an old problem. Pediatr Surg Int. 2001 Sep;17(7):513-4. doi: 10.1007/s003830100584. PMID 11666047